CLINICAL TRIAL: NCT05994417
Title: Objectively Assessed Skin Color and Its Association With Pulse Oximeter Bias in Critically Ill Infants
Brief Title: Beyond Race: Objectively Assessed Skin Color and Its Association With Pulse Oximeter Bias in Critically Ill Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Megha Sharma, Assistant Professor, Section of Neonatology, Department of Pediatrics, University of Arkansas for Medical Sciences, Arkansas Children's Hospital, Arkansas Children's Hospital Research Institute
Other Study IDs: 275653
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Pulse Oximetry; Disparities; Infants
Keywords: pulse oximeter; bias; disparities; infants; premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Arterial blood collected for routine clinical analysis of blood gas status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-Hispanic Black: Infants born to mothers identifying as Non-Hispanic Black
- Non-Hispanic White: Infants born to mothers identifying as Non-Hispanic White
- Infants across the spectrum of melanin index and ITA-based skin color classification

SUMMARY:
The overall objective of this proposal is to quantify the bias in pulse oximeter reported oxygen saturation (SpO2) by evaluating its measures compared to the gold standard blood gas measured arterial oxygen saturation (SaO2) across race and skin pigmentation. The main question that the investigators intend to answer is whether

1. There is greater pulse oximeter bias and subclinical hypoxemia in (1a) Black compared to White infants, and (1b) dark versus light-pigmented infants
2. This bias increases with gestational and postnatal maturation
3. This bias is associated with adverse patient outcomes

DETAILED DESCRIPTION:
The study investigators will conduct a prospective observational study involving 200 infants (0-3 months age) and compare simultaneously obtained pulse oximeter readings (SpO2) and co-oximeter measured blood gas arterial oxygen saturation (SaO2), among infants identified as Non-Hispanic Black and Non-Hispanic White. The investigators will also obtain an objective assessment of skin pigmentation using a non-invasive device, SkinColorCatch® (by Delfin Technologies Ltd, Finland) that provides (1) a melanin index and (2) an objective six-point categorization of skin color based on Individual Typology Angle (ITA). Therefore, the investigators will measure the pulse oximeter bias (SpO2-SaO2) across infants identified as Non-Hispanic Black and Non-Hispanic White, as well as among infants of various skin pigmentation. For infants that have an arterial line for more than one week, the researchers will measure pulse oximeter bias (SpO2-SaO2) on a weekly basis over time with skin maturation and pigmentation changes.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Postnatal age less than 3 months corrected age
* Presence of an in-dwelling umbilical or peripheral arterial line
* Gestational age >= 25 weeks

Exclusion Criteria:

* Known skin pigmentary disorders
* Significantly impaired skin integrity
* Systemic bruising due to birth trauma
* Circulatory shock within last 48 hours
* Infants of peri-viable gestation (22-24 weeks)

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All preterm (i.e. infant less than 37 weeks gestation) and term infants (i.e. infants >= 37 weeks gestation) that have an indwelling arterial line and are admitted to the ACH neonatal intensive care unit (NICU) and cardiovascular intensive care unit (CVICU).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Systematic Bias in pulse oximetry | Within 5 seconds
  The difference between the blood gas measured arterial oxygen saturation (SaO2) and pulse oximeter reported oxygen saturation (SpO2)

SECONDARY OUTCOMES:
Occult Hypoxemia | Within 5 seconds
  The prevalence of occult hypoxemia defined as pulse oximeter reported oxygen saturation (SpO2) of greater than 90% when blood gas measured arterial oxygen saturation (SaO2) is less than 88%.

IPD SHARING:
Plan to Share IPD: Undecided